CLINICAL TRIAL: NCT06662019
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase I Safety Study of Inhaled N-IP-00001 to Determine Tolerability and Safety in Healthy Volunteers.
Brief Title: Phase I Safety Study of Inhaled N-IP-00001 to Determine Tolerability and Safety in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeoTrials Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTPRO-00001
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: safety; tolerability; inhalation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dosing arm (Experimental)
  Interventions: Drug: N-IP-00001 inhalation solution
- Control (Placebo Comparator): Nebulized treatment consisting of 0.9% saline solution.
  Interventions: Drug: 0.9% NaCl isotonic saline solution

INTERVENTIONS:
Drug: N-IP-00001 inhalation solution — Multiple ascending dose (MAD) study. Over the 2 dosing days participants will receive a total of 6 inhaled doses of 5 ml of N-IP-00001 at increasing concentrations, ranging from 0.5mg/ml to 16mg/ml (total volume loaded in the nebuliser is 6 ml per dose).
  Arms: Dosing arm
Drug: 0.9% NaCl isotonic saline solution — Nebulized treatment consisting of 0.9% saline solution.
  Arms: Control

SUMMARY:
Randomized, double-blind, placebo-controlled, dose-escalation Phase I safety study of inhaled N-IP-00001, to determine tolerability and safety in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 55 years.
2. Male or non-pregnant, non-lactating Female
3. Normally active and in good health as determined by the investigator or sub-investigator (who is a qualified physician)through physical examination, vital signs and laboratory parameters.
4. No current acute or chronic respiratory conditions.
5. FEV1 ≥ 80% predicted.
6. Ability to achieve reproducible FEV1 spirometry, as determined by 3 acceptable maneuvres within no more than 5 attempted maneuvres. The best two values should be within 5% or 150mL of each other, whichever is greater.
7. Ability to comply with study medication use, study visits, and study procedures as judged by the investigator.
8. Able to understand and sign an informed consent.
9. Non-smoker and has not smoked for at least 6 months.

Exclusion Criteria:

1. Bowel disease
2. Bariatric surgery
3. Evidence of biliary cirrhosis with portal hypertension
4. History of any drug or alcohol abuse in the past 1 year defined as >21 units of alcohol per week for males and >14 units of alcohol per week for females. Where 1 unit = 360ml of beer, 150ml of wine, or 45ml of spirits.
5. History of lung transplant.
6. History of asthma.
7. History of allergic reactions to fermented foods (kimchi, yoghurt, kefir, kombucha, sauerkraut)
8. Antibiotic treatment within 4 weeks prior to screening
9. Recent (2 weeks) upper respiratory tract infection or COVID
10. Recurrent cough
11. Poor venous access
12. Unexplained, positive drugs of abuse or alcohol breath test results at the screening visit or positive alcohol breath test at check-in.
13. Not able and willing to refrain from alcohol from 24 hours before the first dose through study confinement
14. Unwilling to abstain from fermented foods (kimchi, yoghurt, kefir, kombucha, sauerkraut) and strenuous exercise for 24 hours prior to dosing. Unwilling to abstain from consuming caffeine and/or xanthene products (e.g., coffee, tea, chocolate, and caffeine-containing sodas, colas) during confinement at the clinical unit'.
15. Participants who have received any investigational drug in a clinical research study within the previous 30 days prior to screening or 5 half-lives, whichever is longer.
16. Failure to satisfy the investigator of fitness to participate for any other reason.
17. Currently taking any medication by the inhaled route.
18. Those with commercial interest in the product or related products.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to 2 weeks
FEV1 measured by spirometry | Up to 2 weeks
Changes in vital signs | Up to 2 weeks
  Changes in blood pressure, temperature, pulseoximetry, and heart rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research Ltd, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided